CLINICAL TRIAL: NCT01462734
Title: MicroRNA Expression in Human Blood Serum and Vitreous Body
Status: Completed | Type: Observational
Sponsor: Kyorin University (Other)
Responsible Party: Principal Investigator, Kazunari Hirota, MD, Kyorin University
Other Study IDs: No. 461
Record Dates: First submitted 2011-10-26; First posted 2011-10-31 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: MicroRNA Expression Profile in Human Vitreous
MeSH Terms: interventions — Polymerase Chain Reaction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 3ml of blood serum and 1ml of vitreous
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- human vitreous, human blood serum, PCR: Vitreous and bloodserum samples from macula hole patients without previous ocular or systemic disease
  Interventions: Procedure: human vitreous and blood serum sampling, PCR

INTERVENTIONS:
Procedure: human vitreous and blood serum sampling, PCR — 1ml of human vitreous and 3ml of human blood serum

SUMMARY:
MicroRNAs are important regulators of many cellular functions but their expression profile in human vitreous is still unclear. Aim of this study is to investigate microRNA expression profile by PCR in human vitreous of macula hole patients which is suggested to be similar to that of healthy patients.

ELIGIBILITY:
Inclusion Criteria:

* Female macula hole patients without previous ocular or systemic disease.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Female pateints undergoing vitrectomy for macula hole without previous ocular or systemic disease
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2011-10; Primary Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
MicroRNA expression profile in human vitreous investigated by PCR | 1month

CONTACTS AND LOCATIONS:
Locations (1):
- Kyorin University School Of Medicine, Tokyo, Mitakasi Sinkawa6-20-2, Japan